CLINICAL TRIAL: NCT00050115
Title: Collection of Blood, Stool, Bone Marrow and/or Tissue Samples From Subjects With Hepatitis-Associated Aplastic Anemia
Brief Title: Collection of Biological Samples From Patients With Hepatitis-Associated Aplastic Anemia
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030051; 03-H-0051
Record Dates: First submitted 2002-11-21; First posted 2002-11-20 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis-Associated Aplastic Anemia
Keywords: Bone Marrow Failure; Seronegative Hepatitis; Fulminate Hepatitis; Hepatitis; Aplastic Anemia; Hepatitis Associated Aplastic Anemia
MeSH Terms: conditions — Bone Marrow Failure Disorders; Hepatitis; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatitis A + AA cohort: Subjects seen either at Clinical center or by outside physician

SUMMARY:
This study will collect samples of blood, stool, bone marrow, or other tissues from patients with hepatitis-associated aplastic anemia to investigate a possible association between exposure to viruses and the development of aplastic anemia in these patients. Cells from the samples obtained may be grown in the laboratory for future studies. Patients samples may be used to:

* Study abnormalities that occur in hepatitis-associated aplastic anemia;
* Test for various viruses;
* Test immune function;
* Measure factors related to the patients disease or diseases they may be at risk for;
* Evaluate the effectiveness of current therapies, refine treatment approaches, and identify potential new therapies;
* Identify possible measures for disease prevention;
* Identify possible genetic factors associated with hepatitis-associated aplastic anemia.

Patients 2 years of age and older with severe aplastic anemia that developed within 6 months of an episode of hepatitis may be eligible for this study.

Participants will complete questionnaires and provide tissue samples as described below.

Questionnaires

All patients (or another respondent for the patient) will fill out a questionnaire including demographic information (age, gender, race, ethnic group, education level, state of residence), current symptoms, medications, medical history, and history of possible exposures to toxins or viruses. A second questionnaire, which includes questions related to mental health, sexual behavior, alcohol and drug use, is optional for participants age 21 and older. These questionnaires are designed to uncover features of hepatitis-associated aplastic anemia and possibly reveal a common cause of the disease.

Sample Collections

* Blood- will be collected at the time of the patient s initial evaluation or upon enrollment into the study and possibly periodically during the study. Blood will be drawn through a needle in an arm vein.
* Bone marrow- may be collected as part of the patient s standard medical care or specifically for research purposes of this study. For this procedure, the skin over the hipbone and the outer surface of the bone itself are numbed with an injection of a local anesthesia. Then, a larger needle is inserted into the hipbone and marrow is drawn into a syringe. Marrow cells are suctioned two to six times during the 15-minute procedure.
* Stool- will be provided by the patient.

Liver- tissue may be biopsied as part of the patient s general medical care or for NIH patients, as part of their enrollment in a treatment protocol.

DETAILED DESCRIPTION:
Our laboratory has a long-standing interest in viruses that affect the bone marrow, especially those causing bone marrow failure. One specific syndrome, hepatitis-associated aplastic anemia, suggests that the same agent is responsible for the severe and sometimes fulminate hepatitis as well as the profound bone marrow failure. This study is designed to collect clinical data, and samples from patients with hepatitis-associated aplastic anemia, in order to learn more about the clinical features of the disease, as well as to collect blood, liver, bone marrow and stool samples where possible for ongoing virological studies. For liver and bone marrow samples, material will only be obtained when the liver or bone marrow are biopsied for other medical indications, or during the removal of the liver at the time of transplantation. No additional risk to the patient should result from either procedure.

ELIGIBILITY:
* INCLUSION CRITERIA

Presumptive clinical diagnosis of hepatitis-associated aplastic anemia. That is, aplastic anemia within 12 months of an episode of hepatitis

Age equal to or greater than 2 years old

Ability to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA

Suspected cholestatic or obstructed liver disease

Current diagnosis or past history of myelodysplastic syndrome, Fanconi s anemia, dyskeratosis congenita or other congenital forms of aplastic anemia.

Diagnosis of Diamond-Blackfan anemia or a constitutional marrow failure disease.

Underlying carcinoma, recent history of radiation or chemotherapy

Age less than 2 years old

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2003-03-10 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
to characterize hepatitis disease in subjects with aplastic anemia | Indefinite
  To characterize hepatitis disease in subjects with aplastic anemia

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bottiger LE, Westerholm B. Aplastic anaemia. 3. Aplastic anaemia and infectious hepatitis. Acta Med Scand. 1972 Oct;192(4):323-6. No abstract available. PMID 5081070
- [Background] Mary JY, Baumelou E, Guiguet M. Epidemiology of aplastic anemia in France: a prospective multicentric study. The French Cooperative Group for Epidemiological Study of Aplastic Anemia. Blood. 1990 Apr 15;75(8):1646-53. PMID 2183887
- [Background] Young NS, Issaragrasil S, Chieh CW, Takaku F. Aplastic anaemia in the Orient. Br J Haematol. 1986 Jan;62(1):1-6. doi: 10.1111/j.1365-2141.1986.tb02893.x. No abstract available. PMID 3942690
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-H-0051.html